CLINICAL TRIAL: NCT05736614
Title: Efficacy of a PrEP Uptake & Adherence Intervention Among Male Sex Workers Using a 2-stage Randomization Design
Brief Title: Optimizing PrEP Uptake and Adherence Among Male Sex Workers
Acronym: P4W
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: The Miriam Hospital (Other); University of California, Los Angeles (Other); Project Weber/RENEW (Unknown); Open Door Health (Unknown); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2001002627; R01NR020227 (NIH)
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Prevention
Keywords: PrEP; Prevention; Male Sex Workers (MSW)

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT)
  Study arms:
  1. Stage 1 Standard of Care (SOC) Control Condition
  2. Stage 1 Strength Based Case Management (SBCM) Condition
  3. Stage 2 SOC Control Condition
  4. Stage 2 PrEPare for Work Intervention Condition
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Stage 1 Standard of Care (SOC) Control Condition (No Intervention): SOC participants will receive an informational pamphlet about the PrEP as a form of HIV prevention and referrals to local PrEP Prescribers.
- Stage 1 Strength Based Case Management (SBCM) Condition (Experimental): Intervention participants will receive a trained SBCM to motivate, support, and assist in linkage to PrEP prescribers to help facilitate obtaining PrEP medication to initiate treatment.
  Interventions: Behavioral: Stage 1 Strength Based Case Management (SBCM) Condition
- Stage 2 SOC Control Condition (No Intervention): Research staff will show a brief video that describes what PrEP is and how it works to prevent HIV via sexual and injection transmission. Participants will continue to see their PrEP prescriber for routine clinical care.
- Stage 2 PrEPare for Work Intervention Condition (Experimental): Intervention participants will receive 1-on-1 adherence counseling and personalized daily text messaging reminders to increase PrEP adherence. Intervention participants will undergo three adherence intervention sessions (once per week for 3 weeks) with interventionist.
  Interventions: Behavioral: Stage 2 PrEPare for Work Intervention Condition

INTERVENTIONS:
Behavioral: Stage 1 Strength Based Case Management (SBCM) Condition — Intervention participants will receive a trained SBCM to motivate, support, and assist in linkage to PrEP prescribers to help facilitate obtaining PrEP medication to initiate treatment.
  Arms: Stage 1 Strength Based Case Management (SBCM) Condition
Behavioral: Stage 2 PrEPare for Work Intervention Condition — Intervention participants will receive 1-on-1 adherence counseling and personalized daily text messaging reminders to increase PrEP adherence. Intervention participants will undergo three adherence intervention sessions (once per week for 3 weeks) with interventionist.
  Arms: Stage 2 PrEPare for Work Intervention Condition

SUMMARY:
"PrEPare for Work" is a randomized controlled trial (RCT) whose goal is to test the efficacy of a behavioral intervention (Short Title: PrEPare for Work) in improving PrEP uptake, adherence, and persistence among male sex workers (MSW)

DETAILED DESCRIPTION:
A theory-based, manualized intervention -called "PrEPare for Work"-includes two separate but complementary interventions that address MSW-specific behavioral, economic, interpersonal & structural-level barriers to accessing and adhering to PrEP: 1) peer-led, strengths-based case management (SBCM) for PrEP linkage and uptake; and 2) a technology and counseling intervention to optimize PrEP adherence (once they have access to PrEP). This research will test the PrEPare for Work intervention in a fully-powered RCT to assess efficacy and cost-effectiveness.

ELIGIBILITY:
Inclusion

* Age: 18 years or older
* Assigned male sex at birth
* Identifies as male at enrollment
* Report having engaged in condomless anal sex with another man in the past 3 months
* Report having exchanged sex for money, drugs, items of value, or a place to stay with another man in the past 3 months
* Report HIV status as negative or unsure
* Not currently on PrEP
* Able to understand and speak English or Spanish

Exclusion

* Unable to provide informed consent due to severe mental or physical illness, cognitive impairment, or substance intoxication at the time of interview (will use an adapted version of the Evaluation to Sign Consent Form65 to assess capacity)
* Discovery of active suicidal ideation or major mental illness (e.g. untreated psychosis or mania) at the time of interview (these patients will be referred immediately for treatment)
* Laboratory or clinical findings that would preclude PrEP initiation (e.g. Chronic Hepatitis B Virus infection, decreased creatinine clearance)
* Participated in the pilot RCT and initiated PrEP during study participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological male at birth and current male gender identity
Enrollment: 500 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Stage one: PrEP initiation | 2-month post Stage 1 randomization
  Stage one: PrEP initiation will be measured via verification of prescription filled within two months post-randomization, associated medical records from a PrEP prescriber, and self-report.
Stage two: PrEP adherence | 12-month post Stage 2 randomization
  Stage two: PrEP adherence will be measured via tenofovir concentration in hair. Self-reported adherence will supplement biological monitoring data at 4-month intervals.

SECONDARY OUTCOMES:
PrEP persistence | 12-month post Stage 2 randomization
  PrEP persistence will be measured via medical records and self-report. We will assess PrEP persistence using medical and pharmacy records to confirm provider follow-up visits and prescription refill maintenance. As per Coy et al., PrEP persistence will be defined as having ≥16 days of PrEP medication filled per 30-day period, for at least three-quarters of the months since initiation to study completion (~9 months).

CONTACTS AND LOCATIONS:
Overall Officials: Katie Biello, PhD, Principal Investigator — Brown University School of Public Health
Locations (5):
- United States (5):
  - UCLA Fielding School of Public Health, Los Angeles, California
  - The Miriam Hospital, Providence, Rhode Island
  - Open Door Health, Providence, Rhode Island
  - Project Weber/RENEW, Providence, Rhode Island
  - Brown University School of Public Health, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that this data will be presented annually on data collected after the second year when sufficient baseline data is collected. It is anticipated that most of the papers and data-based projects/presentations will happen in year 3, when all of the baseline data is collected, and the 3 month outcome has occurred for all participants. Sharing of the findings will involve a primary paper describing the study outcome and a paper that describes the intervention, as well as submitting to lead workshops on the intervention approach at relevant national meetings and conferences. Raw data for additional analysis will be available to outside individuals through contacting the MPIs. Information regarding the availability of data for analysis will be listed on the MPIs' web pages. Contact information for the MPIs will be listed in all manuscripts and publications as another means to access data.
Supporting Information: Study Protocol
Time Frame: Raw data for additional analysis will be available to outside individuals through contacting the MPIs at two different times. The first will be after all of the baseline data is collected. The second will be after the publication and release of the primary outcome paper(s). The MPIs will store the data indefinitely and allow access for pooled data analysis projects, or projects for outside individuals.
Access Criteria: Raw data for additional analysis will be available to outside individuals through contacting the MPIs. We will institute a concept plan process where internal study staff first have the availability to write papers or give presentations on particular topics. After this, if outside individuals wish to analyze data, we will welcome this collaboration.

REFERENCES:
- [Derived] Biello KB, Chan PA, Ndoye CD, Nelson L, Nelson E, Silva V, Kwak E, Napoleon S, Cormack Orellana C, Richards OG, Davis E, Mimiaga MJ. Study protocol of a randomized controlled trial to assess the efficacy of the "PrEPare for Work" intervention to enhance PrEP uptake and optimize adherence for HIV prevention among male sex workers in the U.S. BMC Public Health. 2024 Feb 9;24(1):424. doi: 10.1186/s12889-024-17710-y. PMID 38336731